CLINICAL TRIAL: NCT01756248
Title: Special Drug Use Investigation of EYLEA for AMD
Brief Title: EYLEA Age-Related Macular Degeneration (AMD) Post-marketing Surveillance in Japan
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Collaborators: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Other Study IDs: 15895; EYL-AMD (Other: company internal)
Record Dates: First submitted 2012-12-20; First posted 2012-12-25 (Estimated); Last update posted 2023-06-07 (Actual); Status verified 2023-06

CONDITIONS: Macular Degeneration
Keywords: EYLEA; Age-Related Macular Degeneration
MeSH Terms: conditions — Macular Degeneration | interventions — aflibercept

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Group 1
  Interventions: Drug: Aflibercept(Eylea, VEGF Trap-Eye, BAY86-5321)

INTERVENTIONS:
Drug: Aflibercept(Eylea, VEGF Trap-Eye, BAY86-5321) — Patients treated with EYLEA under practical manner for AMD.

SUMMARY:
This study is a regulatory post-marketing surveillance in Japan, and it is a local prospective and observational study of patients who have received EYLEA for Age-Related Macular Degeneration (AMD).

The objective of this study is to assess safety and effectiveness of EYLEA using in real clinical practice.

A total of 4,000 patients are to be enrolled and assessed in 3 years standard observational period. An annual follow-up survey will be conducted for 5 years at the longest after standard observational period.

ELIGIBILITY:
Inclusion Criteria:

* Patients who received EYLEA for AMD

Exclusion Criteria:

* Patients who have already received EYLEA

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with subfovear choroidal neovascular age-related macular degeneration
Sampling Method: Non-Probability Sample
Enrollment: 3872 (Actual)
Dates: Start 2012-12-26 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2019-05-20 (Actual)

PRIMARY OUTCOMES:
Number of participants with adverse drug reactions(ADRs) and infections from the first intravitreal(ITV) injection of EYLEA | Up to 3 years
Number of participants with serious adverse events (SAEs) and ocular adverse events(AEs) (especially AEs due to ITV injection procedure) from the first ITV injection of EYLEA | Up to 3 years

SECONDARY OUTCOMES:
Number of participants with ADRs, SAEs and ocular AEs ( especially AEs due to ITV injection procedure) in subpopulations of patients background characteristics and status of EYLEA treatments from the first ITV injection of EYLEA | Up to 3 years
Mean changes in visual acuity | Baseline and 6, 24 or 36 months
Proportion of patients who maintained visual acuity(corresponding to <15 letters of Early Treatment Diabetic Retinopathy Study(ETDRS) from baseline) and improved visual acuity(corresponding to >0 letter of ETDRS from baseline) | Up to 3 years
Mean changes in visual acuity in subpopulations of patients background characteristics and status of EYLEA treatments | Baseline and 6, 24 or 36 months
Number and intervals of ITV injection of EYLEA | Up to 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- Multiple Locations, Japan

REFERENCES:
- [Derived] Ozawa Y, Ohgami K, Sasaki K, Hirano K, Sunaya T. Long-term surveillance provides real-world evidences of safety and effectiveness in intravitreal aflibercept treatment for age-related macular degeneration. Sci Rep. 2023 Jun 30;13(1):10597. doi: 10.1038/s41598-023-37584-1. PMID 37391547
- See also: Click here to find information for studies related to Bayer products. To find this study enter the ClinicalTrials.gov identifier (NCT) number or Bayer Study Identifier (ID) in the search field — http://clinicaltrials.bayer.com/